CLINICAL TRIAL: NCT04934787
Title: Exo-neuro-musculo-skeleton With Balance Sensing Feedback for Ankle-foot Rehabilitation After Stroke
Brief Title: ENMS With Balance Feedback for Post-stroke Ankle-foot Rehabilitation
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Hong Kong Polytechnic University (Other)
Collaborators: Innovation and Technology Commission, Hong Kong (Other); Prince of Wales Hospital, Shatin, Hong Kong (Other)
Responsible Party: Principal Investigator, Xiaoling Hu, Assistant Profession, The Hong Kong Polytechnic University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ITS/062/19
Record Dates: First submitted 2021-06-03; First posted 2021-06-22 (Actual); Last update posted 2025-04-08 (Actual); Status verified 2025-04

CONDITIONS: Cerebrovascular Stroke; Foot Drop; Foot Inversion Deformity
Keywords: Robot; Stroke; Lower limb
MeSH Terms: conditions — Stroke; Peroneal Neuropathies

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- ENMS-BSF assisted gait training (Experimental): The participants will receive the full assistance of the ENMS-BSF during a 20-session gait rehabilitation.
  Interventions: Device: ENMS-BSF assisted gait training
- Partial ENMS-BSF assisted gait training (Active Comparator): The participants will receive a partial assistance of the ENMS-BSF during a 20-session gait rehabilitation.
  Interventions: Device: ENMS-BSF assisted gait training
- Sham ENMS-BSF assisted gait training (Sham Comparator): The participants will only wear the device without assistance during a 20-session gait rehabilitation.
  Interventions: Device: ENMS-BSF assisted gait training

INTERVENTIONS:
Device: ENMS-BSF assisted gait training — 1. ENMS-BSF will correct the foot-drop and foot inversion during post-stroke walking.
  2. Each participant will receive 20 sessions device assisted training, with an intensity of 3-5 sessions/week, 1 hr/session.
  3. In each session, a participant will complete the device-assisted walking on flat ground with a natural speed and with the aid of a four-pronged cane.

SUMMARY:
In this work, a novel hybrid ankle-foot robot is designed for gait rehabilitation after stroke, i.e., exoneuromusculoskeleton with balance sensing feedback (ENMS-BSF) by integrating the advantages of soft pneumatic muscle, functional electrical stimulation, exoskeleton and foot balance feedback in one system. With the assistance of the ENMS-BSF the foot drop and foot inversion could be corrected with improved muscle coordination in the paretic lower limb. The device is wearable and light-in-weight for unilateral application during walking. It is hypothesized that with the intervention of the ENMS-BSF the gait pattern of persons after stroke can be improved with long-term rehabilitative effects.

ELIGIBILITY:
Inclusion Criteria:

* At least 6 months after the onset of stroke
* Have sufficient cognition to follow simple instructions, as well as understand the content and purpose of the experiment (Mini-Mental State Examination (MMSE) score >21).
* Have mild-to-moderate motor impairment in the affected lower limb with foot drop but be capable of standing and walking without manual assistance.
* Fugl-Meyer Assessment (FMA), total score on the lower limb <20
* Functional Ambulatory Category (FAC) ≥4
* Berg Balance Scale (BBS) ≥40

Exclusion Criteria:

* The exclusion criteria will be server spasticity at the ankle joint measured by Modified Ashworth Score (MAS) >3.
* Receiving other lower limb rehabilitative interventions at the same time

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2021-07-01 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Change in Fugl-Meyer Assessment | before, one day after, and 3 months after the training
  To evaluate the voluntary motor function of the lower limb after the interventions

CONTACTS AND LOCATIONS:
Locations (1):
- The Hong Kong Polytechnic University, Hong Kong, China

IPD SHARING:
Plan to Share IPD: No
According to the obtained ethical approval, all personal data of participants cannot be shared or released.